CLINICAL TRIAL: NCT02542826
Title: Constant Rate Shuttle Walking and Stair Stepping Tests to Assess Exertional Dyspnea in COPD: Responsiveness to Pulmonary Rehabilitation and Minimal Clinically Important Difference
Brief Title: Pulmonary Rehab, Dyspnea, Walk and Step Testing in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Mount Sinai Hospital, Montreal (Other); Laval University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-CUSM-15-074
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Rehabilitation; 3-minute constant rate shuttle walk test; 3-minute constant rate step test; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental)
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Patients will participate in 3 exercise training sessions/wk for a period of 7-12 wks at one of 4 sites in Quebec. Each training session will include 30-45 min of aerobic training (cycling and/or treadmill walking) at a target intensity of 80% of the maximal heart rate achieved during a symptom-limited incremental cycle exercise test performed prior to the pulmonary rehabilitation program; and 20-30 min of strength training exercises.

SUMMARY:
This is a multi-site collaborative study that will be done in the context of three Quebec hospitals' outpatient pulmonary rehabilitation programs: Montreal Chest Institute; University of Laval, and Hopital Sacre-Coeur Montreal. The objectives are two-fold. First, to determine the Minimal Clinical Important Difference in intensity ratings of perceived breathlessness for each of the 3-min constant rate shuttle walking (3-MWT) and stair stepping (3-MST) protocols in patients with chronic obstructive pulmonary disease (COPD). Second, to test the hypothesis that both the 3-MWT and 3-MST protocols are able to detect statistically significant and clinically-meaningful improvements in exertional breathlessness following an 7-12 week outpatient rehabilitative exercise training program in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ambulatory
* Moderate-to-very severe COPD (GOLD Stage 2-4)

Exclusion Criteria:

* Respiratory exacerbation in the previous 6 weeks
* Change in medication dosage/frequency in the previous 6 weeks
* Clinical evidence of asthma
* Cardiovascular and/or neuromuscular diseases that are unstable and/or that may contribute to exercise limitation
* Any other contraindications to exercise training/testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-04 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Minimal clinically important difference (MCID) with regards to the change in breathlessness intensity ratings at the end of each of the 3-MST and 3-MWT. | Baseline and 7 weeks

SECONDARY OUTCOMES:
Change (post- minus pre- pulmonary rehab) in dyspnea intensity ratings on the Borg 0-10 ratio category scale | Baseline and 7 weeks
  Borg 0-10 category ratio scale

OTHER OUTCOMES:
Change (post- minus pre- pulmonary rehab) in spirometry (FEV1, FVC, and FEV1/FVC) | Baseline and 7 weeks
  expressed in L and as % predicted
Change (post- minus pre- pulmonary rehab) in lung volumes (TLC, FRC, RV) | Baseline and 7 weeks
  expressed in L and as % predicted
Change (post- minus pre- pulmonary rehab) in airways resistance (Raw, sRaw) | Baseline and 7 weeks
  expressed in L and as % predicted
Change (post- minus pre- pulmonary rehab) CCQ | Baseline and 7 weeks
  questionnaire
Change (post- minus pre- pulmonary rehab) CRQ | Baseline and 7 weeks
  questionnaire
Change (post- minus pre- pulmonary rehab) IPAQ | Baseline and 7 weeks
  questionnaire
Change (post- minus pre- pulmonary rehab) BDI/TDI | Baseline and 7 weeks
  questionnaire
Change (post- minus pre- pulmonary rehab) CAT | Baseline and 7 weeks
  questionnaire
Change (post- minus pre- pulmonary rehab) in Exercise Endurance Time (EET) to constant power output cycling exercise performed at 75% of the peak incremental cycling power output achieved prior to start of pulmonary rehab | Baseline and 7 weeks
  EET, in minutes and sec
Change (post- minus pre- pulmonary rehab) in peak VO2 to constant power output cycling exercise performed at 75% of the peak incremental cycling power output achieved prior to start of pulmonary rehab | Baseline and 7 weeks
  in ml/kg/min and as %predicted
Change (post- minus pre- pulmonary rehab) in peak Ventilation to constant power output cycling exercise performed at 75% of the peak incremental cycling power output achieved prior to start of pulmonary rehab | Baseline and 7 weeks
  in L/min, as %predicted and as % of MVV (=FEV1x35)
Change (post- minus pre- pulmonary rehab) in the 6-minute walk distance | Baseline and 7 weeks
  in m
Change (post- minus pre- pulmonary rehab) in body composition assessed by dual-energy X-ray absorptiometry | Baseline and 7 weeks
  Lean body mass (g)
Change (post- minus pre- pulmonary rehab) in isometric quadriceps peak torque | Baseline and 7 weeks
  % predicted

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- McConnell Centre for Innovative Medicine, Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl/